CLINICAL TRIAL: NCT03516370
Title: Effect Of A Locally Delivered Probiotic Sacchraomyces Boulardii As An Adjunct To Scaling And Root Planing In The Management Of Chronic Periodontitis: A Randomized, Split Mouth, Single Blind, Clinico-Microbiological Study
Brief Title: Effect Of A Locally Delivered Probiotic Sacchraomyces Boulardii In The Management Of Chronic Periodontitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tatyasaheb Kore Dental College (Other)
Responsible Party: Principal Investigator, Dr.Kshitij .K. Karmkar, Principle investigator, Tatyasaheb Kore Dental College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 9403303401
Record Dates: First submitted 2018-04-26; First posted 2018-05-04 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Chronic Periodontitis
Keywords: chronic periodontitis; Sacchraomyces boulardii; probiotics
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant
Masking Description: patients were masked they didnt know which mixture they recived during treatment ensuring single blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Scaling and root planning was followed by placement of Lyophilized Saccharomyces Boulardii 250 MG in the pocket. S. boulardii was delivered subgingivally by by mixing 1gm of sachet containing 250mg of lyophilized yeast with 0.5ml of distilled water this prepared paste was injected in the perio pocket with luer lock syring and cannula.
  Interventions: Drug: Saccharomyces Boulardii 250 MG
- control group (Placebo Comparator): Control site received placebo i.e distilled water as a mixture after scaling and root planning.
  Interventions: Drug: Saccharomyces Boulardii 250 MG

INTERVENTIONS:
Drug: Saccharomyces Boulardii 250 MG — all the patient first recived scaling and root planning as a prophylactic mesaure later after that patient received intrapocket delivery of Saccharomyces Boulardii mixture.
  Other Names: scaling and root planning

SUMMARY:
This study was carried out in the Department of Periodontology and source of patient was be from the outpatient section of Tatyasaheb Kore Dental College & Research Centre, New Pargaon. Study included the 31 patients with chronic periodontitis, with age group between 35-60 years, two interdental suprabony pockets with 5-8mm pocket depth in two different quadrants were chosen as the test site (TS) and control sites (CS). In control sites, only SRP was performed followed by placement of placebo distilled water. In test sites, SRP was followed by placement of Lyophilized saccharomyces boulardii in the pocket. S. boulardii will be delivered subgingivally by by mixing 1gm of sachet containing 250mg of lyophilized yeast with 0.5ml of distilled water this prepared paste was injected in the perio pocket with luer lock syringe and cannula .The subgingival plaque samples were collected at baseline, 4th day, 4 week for detection of p. gingivalis for microbiological analysis and clinical parameters wiere recorded at baseline and at 1 month.

DETAILED DESCRIPTION:
1. AIM: To determine effectiveness of saccharomyces boulardii as an adjuvant to scaling and root planing in the treatment of chronic periodontitis 2. OBJECTIVES:

1. To evaluate the efficacy of locally delivered saccharomyces boulardii on clinical and microbiological parameters in the treatment of chronic periodontitis.
2. To compare the result of scaling and root planning alone and scaling and root planing with locally delivered saccharomyces boulardii in patients with chronic periodontitis.

MATERIALS AND METHODS:- A split mouth, single blind, randomized placebo controlled, clinical & microbiologic study was carried out in 31 patients at the department of Periodontology. Based on power of study i.e 95% and with alpha (α )of 0.05 the sample size finalized was 31. Prior approval for the study was obtained from the Local Ethical Committee. Two interdental suprabony pockets with 5-8mm pocket depth in two different quadrants were chosen as the test site (TS) and control sites (CS).

CONSENT After the study was explained, including the benefits, risks, and alternative treatments, the patients signed an informed consent form indicating their agreement to participate in the study, and each patient was assigned a patient number in ascending order to maintain the masking of evaluators. Eg. First patient was given a number D1, Second D2, and so on.

GROUPS This was a Phase 2 clinical trial with an Interventional model of parallel assignment with two arms. Hence, after screening through inclusion and exclusion criteria in single patient two sites were selected in contralateral quadrants through randomization. 31sites were included in test site and 31 sites were included in control site.

Test Site (TS):- SRP was followed by placement of Lyophilized S boulardii in the pocket. S. boulardii was delivered subgingivally by by mixing 1gm of sachet containing 250mg of lyophilized yeast with 0.5ml of distilled water this prepared paste was injected in the perio pocket with luer lock syring and cannula. Periodontal pack was given in delivered area to maintain the mixture into the pocket and patients were advised not to brush in that area. A stent was prepared and probing pocket depth was measured before and after the treatment. The stent enabled the periodontal probe to reach the same position before and after the treatment, to avoid error or bias during treatment.

Control Site (CS):- Control site received placebo i.e distilled water after scaling and root planning.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy subject.
2. Presence of minimum 16 teeth.
3. Patient with generalized moderate to severe chronic periodontitis.
4. Probing depth (PD) 5-8mm.
5. Clinical Attachment Level > 4mm

Exclusion Criteria:

1. Tobacco in any form and alcoholics.
2. Pregnant and lactating mother.
3. Patients with history of systemic ailments, patients under ant-inflammatory/antibiotic/antifungal/probiotic/prebiotic 6 months prior to recruitment for study.
4. Subjects who had received periodontal treatment within the previous 6 months.
5. Aggressive periodontitis.
6. Patients with confirmed or suspected intolerance to S,boulardii derivatives will be excluded from the study.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
pocket depth reduction | 1 month
  after subgingival delivery of lyophilized s. boulardi mixture the pocket depth shiuld recived after 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Dilip Khambete, MDS, Study Chair — tatayasaheb kore dental college and hospital new pargaon
Locations (1):
- Dental, Kolhāpur, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided